CLINICAL TRIAL: NCT00910650
Title: Adoptive Transfer of MART-1 F5 TCR Engineered Peripheral Blood Mononuclear Cells (PBMC) After a Nonmyeloablative Conditioning Regimen, With Administration of MART-126•35-Pulsed Dendritic Cells and Interleukin-2, in Patients With Advanced Melanoma
Brief Title: Study of Gene Modified Immune Cells in Patients With Advanced Melanoma
Acronym: F5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: California Institute of Technology (Other); University of Southern California (Other); University of Connecticut (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-001212; 08-02-020 (Other: UCLA IRB)
Record Dates: First submitted 2009-05-01; First posted 2009-06-01 (Estimated); Results first posted 2021-08-04 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2020-02

CONDITIONS: Metastatic Melanoma
Keywords: Adoptive transfer therapy; Dendritic cell vaccines
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F5 TCR transgenic cells (Experimental): F5 TCR transgenic cell adoptive transfer therapy
  Interventions: Biological: F5 TCR transgenic cells and MART-1 peptide pulsed dendritic cells; Drug: non-myeloablative conditioning chemotherapy

INTERVENTIONS:
Biological: F5 TCR transgenic cells and MART-1 peptide pulsed dendritic cells — After chemotherapy, patients receive up to 1 x 10(9) MART-1 F5 TCR transgenic T cells infused i.v., 1 x 10(7) MART-1 peptide pulsed dendritic cells intradermally, and low dose IL-2 500,000 IU/m2 s.c. twice daily for 14 days.
  Other Names: F5 TCR transgenic cells; MART-1 peptide pulsed dendritic cells; Interleukin-2 (aldesleukin)
Drug: non-myeloablative conditioning chemotherapy — Patients receive non-myeloablative conditioning chemotherapy with Cyclophosphamide 60 mg/kg/day x 2 days and Fludarabine 25 mg/m2/day i.v. over 30 minutes for 4 days

SUMMARY:
The purpose of this phase 2 study is to find the best way to give this new experimental regimen and determine if it can treat metastatic melanoma in humans. In this phase 2 study, the experimental products are given initially to a group of 8 people. If safe and found to have significant anti-tumor activity, it will be given to up to 14 other people, for a total of 22 people in this study. Physicians watch subjects carefully for any harmful side effects. Although the experimental regimen has been well tested in laboratory and animal studies, and a similar regimen has been given to a group of patients at the National Cancer Institute in Bethesda, MD, the side effects in people cannot be completely known ahead of time. This protocol is offered only to people whose condition cannot be helped by other known treatments.

The study procedures will start with the collection of white blood cells through apheresis (a procedure in which blood is drawn from a patient and separated into its components, some of which are retained, such as white blood cells, and the remainder returned by transfusion to the patient).

Subjects will be asked to undergo two aphereses, one to make the gene-modified MART-1 TCR CTLs (cytolytic T lymphocyte) and the dendritic cell vaccines, and a second one after the subject receives the gene modified cells to later study them in the blood.

On the day of the first apheresis, subjects will be admitted to the hospital and will receive chemotherapy over the next five days which decreases the risk of rejection of the transferred cells by the subject's immune system and facilitates their expansion and attack of the melanoma lesions. During this time, the gene-modified MART-1 TCR CTLs and the dendritic cells will be manufactured in the laboratory from the apheresis product and will be extensively tested to assure that they express the appropriate TCR and that they do not contain any contaminating bacteria or virus. Then the gene-modified MART-1 TCR CTLs will be given back to the subject through a vein in the arm. It will be followed by vaccination with the dendritic cells under the skin. During the next fourteen days, subjects will also receive interleukin 2 (IL-2), which is a standard treatment for patients with metastatic melanoma. During the next 2 to 3 weeks, subjects will stay in the hospital until the study investigators determine that the subject has fully recovered from all of the procedures, and it is safe for the subject to go home. Chemotherapy frequently causes a decrease in the platelet or red blood cells, and therefore subjects may require platelet and/or red blood cell transfusions.

DETAILED DESCRIPTION:
This is a two-stage phase II clinical trial with the combined primary endpoints to determine the safety, feasibility and anti-tumor activity of adoptive transfer of peripheral blood mononuclear cells (PBMC) genetically engineered to express the alpha and beta chains of a high affinity T cell receptor (TCR) specific for the HLA-A*0201-restricted MART-1 melanoma tumor antigen to patients with locally advanced or metastatic melanoma. This gene transfer will be facilitated by a retroviral vector pseudotyped with a gibbon ape leukemia virus (GaLV) envelope. The two transgenes are linked by a picornavirus 2A sequence. Their expression is driven by the retroviral long terminal repeat (LTR).

Patients with MART-1-positive locally advanced or metastatic melanoma who are HLA-A*0201-positive, and HIV, hepatitis B and C seronegative, will receive a non-myeloablative but lymphocyte depleting chemotherapy conditioning regimen consisting of cyclophosphamide and fludarabine, and then receive the adoptive transfer of autologous PBMC transduced with the MSGV1-F5AfT2AB retroviral vector, which expresses a high affinity TCR for the MART-1 melanoma antigen (MART-1 F5 TCR). The cell dose will be up to 10^9 autologous PBMC transduced with the MSGV1-F5AfT2AB retroviral vector. The transgenic T cells will be infused fresh on the day of harvest as done in the last three patients within this protocol, prior to which, thawed cryopreserved cells were infused. Following adoptive cell transfer, patients will receive MART-1.26-35 peptide-pulsed dendritic cell (DC) vaccines and low dose interleukin-2 (IL-2).

The MART-1 F5 TCR was provided by Dr. Stephen A. Rosenberg from the Surgery Branch, National Cancer Institute (NCI). The MART-1 F5 TCR is derived from the DMF5 tumor infiltrating lymphocyte (TIL) clone, and was selected from several MART-1-specific TCRs because of its high affinity and biological activity. This TCR delivered by the same retroviral vector is currently in clinical testing at the Surgery Branch/NCI. Both the NCI clinical trial and the trial at University of California at Los Angeles (UCLA) are based on the same retrovirus expressing the MART-1 F5 TCR used to transduce whole PBMC and re-infused to patients after a non-myeloablative but lymphodepleting chemotherapy conditioning regimen. Major differences between both clinical trials include the shorter ex vivo expansion of TCR transduced PBMC, the use of MART-126-35 peptide pulsed DC and the use of positron imaging tomography (PET) for non-invasive imaging of adoptively transferred TCR transgenic cells in the UCLA clinical trial.

The primary endpoints will be safety, feasibility and objective tumor response. The phase II clinical trial design will have two treatment stages following a Simon optimal two-stage clinical phase II clinical trial design 1. The clinical trial will have an initial stage with 8 patients followed by a second stage with up to 22 patients.

Safety will be determined in stage one, and if 3 out of 8 patients have MART-1 F5 TCR-induced dose limiting toxicities (DLT), then further accrual will not be warranted. Feasibility will be also determined in the first stage, and if 3 out of 8 patients cannot receive the intended cellular therapies, or if they result in suboptimal TCR transgenic cell in vivo persistence, further accrual will not be warranted to the protocol as currently designed. Objective tumor responses will be determined by RECIST objective response criteria with a design to rule out a 10% response rate as the null hypothesis, and a 35% response rate as the alternative hypothesis. With this statistical design, if 2 or more of 8 patients in stage one have an objective response, the study will proceed to stage two and accrue a total of 22 patients. If 5 or more patients in the overall study have a complete response (CR) or partial response (PR), which combined result in the objective response rate, the study will be declared positive.

Secondary study endpoints are transgenic T cell persistence in humans and their ability to home to MART-1 positive melanoma metastasis. Analysis will be performed by sampling of peripheral blood and tumor deposits for T cell persistence and by non-invasive metabolic imaging using PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma that is considered surgically incurable with either:

  * Stage IIIc melanoma including locally relapsed, satellite, in-transit lesions or bulky draining node metastasis.
  * Stage IV melanoma (M1a, M1b or M1c). At least 1 lesion amenable for outpatient biopsies; this should be a cutaneous or palpable metastatic site or a deeper site accessible by image-guided biopsy that is deemed safe to access by the treating physicians and interventional radiologists. Patients without accessible lesions for biopsy but with prior tissue available from metastatic disease would be eligible at the investigator's discretion.
* MART-1 positive melanoma by RT-PCR or Immuno-histochemical (IHC).
* HLA-A*0201 (HLA-A2.1) positivity by molecular subtyping*.
* Age greater than or equal to 18 years old.
* Life expectancy greater than 3 months assessed by a study physician.
* A minimum of one measurable lesion defined as:

  * Meeting the criteria for measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST).
  * Skin lesion(s) selected as non-completely biopsied target lesion(s) that can be accurately measured and recorded by color photography with a ruler to document the size of the target lesion(s).
* No restriction based on prior treatments.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Adequate bone marrow and hepatic function determined within 30-60 days prior to enrollment, defined as:

  * Absolute neutrophil count >= 1.5 x 109 cells/L.
  * Platelets >= 100 x 109/L.
  * Hemoglobin >= 10 g/dL.
  * Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x ULN (=< 5 x ULN, if documented liver metastases are present).
  * Total bilirubin =< 2 x Upper Limit of Normal (ULN) (except patients with documented Gilbert's syndrome).
  * Creatinine < 2 mg/dl (or a glomerular filtration rate > 60).
  * Must be willing and able to accept at least two leukapheresis procedures.
  * Must be willing and able to accept at least two tumor biopsies.
  * Must be willing and able to provide written informed consent.
* Patients with HLA-A*0205 (HLA-A2.5) positivity by molecular subtyping may be eligible if there is demonstration that they can correctly present the MART-126-35 epitope as stimulators for IFN-gamma production by MART-1 F5 TCR transgenic cells.

Exclusion Criteria

* Previously known hypersensitivity to any of the agents used in this study.
* Received systemic treatment for cancer, including immunotherapy, within one month prior to initiation of dosing within this protocol. However, cell harvesting by leukapheresis may be performed before one month from prior therapy if the study investigators consider that it will not have a detrimental impact on the generation of the two cell therapies in this protocol.
* History of, or significant evidence of risk for, chronic inflammatory or autoimmune disease (eg, Addison's disease, multiple sclerosis, Graves disease, Hashimoto's thyroiditis, inflammatory bowel disease, psoriasis, rheumatoid arthritis, systemic lupus erythematosus, hypophysitis, pituitary disorders, etc.). Patients will be eligible if prior autoimmune disease is not deemed to be active (e.g. fibrotic damage of the thyroid after thyroiditis or its treatment, with stable thyroid hormone replacement therapy). Vitiligo will not be a basis for exclusion.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea or bleeding, or current acute colitis of any origin.
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or received systemic steroids within the last 4 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed).
* HIV seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist.
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the chemotherapy conditioning regimen and supportive treatments. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Clinically active brain metastases. Radiological documentation of absence of active brain metastases at screening is required for all patients. Prior evidence of brain metastasis successfully treated with surgery or radiation therapy will not be exclusion for participation as long as they are deemed under control at the time of study enrollment.
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal for two years, or must agree to use effective contraception during the period of treatment and 6 months after. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) within 14 days from starting the conditioning chemotherapy. The definition of effective contraception will be based on the judgment of the study investigators.
* Since IL-2 is administered following cell infusion:

  * Patients will be excluded if they have a history of clinically significant ECG abnormalities, symptoms of cardiac ischemia or arrhythmias and have a left ventricular ejection fraction (LVEF) < 45% on a cardiac stress test (stress thallium, stress MUGA, dobutamine echocardiogram, or other stress test).
  * Similarly, patients who are 50 years old with a baseline LVEF < 45% will be excluded.
  * Patients with ECG results of any conduction delays (PR interval >200ms, QTC > 480ms), sinus bradycardia (resting heart rate <50 beats per minute), sinus tachycardia (HR>120 beats per minute) will be evaluated by a cardiologist prior to starting the trial. Patients with any arrhythmias, including atrial fibrillation/atrial flutter, excessive ectopy (defined as >20 PVCs per minute), ventricular tachycardia, 3rd degree heart block will be excluded from the study unless cleared by a cardiologist.
  * Patients with pulmonary function test abnormalities as evidenced by a forced expiratory volume at one second/forced vital capacity (FEV1/FVC)< 70% of predicted for normality will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10-13 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Principal Investigator — University of California, Los Angeles; Bartosz Chmielowski, MD, PhD, Principal Investigator — University of California, Los Angeles; James S Economou, MD, PhD, Principal Investigator — University of California, Los Angeles; John A Glaspy, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, David Geffen School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Derived] Mehta A, Kim YJ, Robert L, Tsoi J, Comin-Anduix B, Berent-Maoz B, Cochran AJ, Economou JS, Tumeh PC, Puig-Saus C, Ribas A. Immunotherapy Resistance by Inflammation-Induced Dedifferentiation. Cancer Discov. 2018 Aug;8(8):935-943. doi: 10.1158/2159-8290.CD-17-1178. Epub 2018 Jun 13. PMID 29899062
- [Derived] Nowicki TS, Escuin-Ordinas H, Avramis E, Chmielowski B, Chodon T, Berent-Maoz B, Wang X, Kaplan-Lefko P, Yang L, Baltimore D, Economou JS, Ribas A, Comin-Anduix B. Characterization of Postinfusion Phenotypic Differences in Fresh Versus Cryopreserved TCR Engineered Adoptive Cell Therapy Products. J Immunother. 2018 Jun;41(5):248-259. doi: 10.1097/CJI.0000000000000216. PMID 29470191
- [Derived] Ma C, Cheung AF, Chodon T, Koya RC, Wu Z, Ng C, Avramis E, Cochran AJ, Witte ON, Baltimore D, Chmielowski B, Economou JS, Comin-Anduix B, Ribas A, Heath JR. Multifunctional T-cell analyses to study response and progression in adoptive cell transfer immunotherapy. Cancer Discov. 2013 Apr;3(4):418-29. doi: 10.1158/2159-8290.CD-12-0383. Epub 2013 Mar 21. PMID 23519018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 10/13/2009 to 04/04/2013 (suspended); 10/16/2013 to 02/07/2018 (closed for accrual). Location: University of California at Los Angeles medical Clinic.
Groups:
- F5 T-cell Receptor (TCR) Transgenic Cells: F5 TCR transgenic cell adoptive transfer therapy
  F5 TCR transgenic cells and Melanoma antigen recognized by T-cells (MART-1) peptide pulsed dendritic cells: After chemotherapy, patients receive up to 1 x 10(9) MART-1 F5 TCR transgenic T cells infused i.v., 1 x 10(7) MART-1 peptide pulsed dendritic cells intradermally, and low dose Interleukin-2 (IL-2) 500,000 IU/m2 s.c. twice daily for 14 days.
  non-myeloablative conditioning chemotherapy: Patients receive non-myeloablative conditioning chemotherapy with Cyclophosphamide 60 mg/kg/day x 2 days and Fludarabine 25 mg/m2/day i.v. over 30 minutes for 4 days
Period: Overall Study
Arm/Group | F5 T-cell Receptor (TCR) Transgenic Cells
Started | 14
Completed | 12
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | F5 TCR Transgenic Cells
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Response Rate: The Number of Participants Who Completed the Maximum Time Allowed on Study Without Being Affected by Tumor Recurrence or Progression.
Time Frame: every 90 days for up to 3 years
Population: Maximum time in study: 3 years from 1st study drug administration.
Measure: Count of Participants; unit: Participants
Arm/Group | F5 TCR Transgenic Cells
Number analyzed (Participants) | 14
Participants | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is measured until the patient passes away
Time Frame: Baseline from treatment for the life of the participant > 7 years
Measure: Count of Participants; unit: Participants
Arm/Group | F5 TCR Transgenic Cells
Number analyzed (Participants) | 14
Participants
  Deceased | 14
  Alive | 0

ADVERSE EVENTS:
Time Frame: 3 months and 1 week
Description: Adverse Events and Serious Adverse Events monitored for the treatment period, 3 months and 1 week.
  All Cause mortality accessed for balance of participants life, up to seven years.
Arm/Group | F5 TCR Transgenic Cells
All-Cause Mortality (participants affected / at risk) | 14/14
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F5 TCR Transgenic Cells (N=14)
Anemia (Vascular disorders) | 2 (2)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Deep Vein Thrombosis left subclavian (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Pancytopenia (Cardiac disorders) | 1 (1)
Rapid Drop in Hemoglobin level (Cardiac disorders) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 2 (2)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Seizures (Nervous system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F5 TCR Transgenic Cells (N=14)
Abdomen distention (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal fullness (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abnormal Urinalysis (Renal and urinary disorders) | 2 (2)
Acidemia (Cardiac disorders) | 1 (1)
Agitation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline Phosphate Level elevated (Cardiac disorders) | 4 (4)
Alopecia (Musculoskeletal and connective tissue disorders) | 1 (1)
Altered level of consciousness (Psychiatric disorders) | 1 (1)
Anasarca (Musculoskeletal and connective tissue disorders) | 1 (1)
absolute neutrophil count (Cardiac disorders) | 2 (2)
Anemia (Cardiac disorders) | 11 (11)
Anorexia (Gastrointestinal disorders) | 4 (4)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspartate Aminotransferase increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Atrial fibrilation (Cardiac disorders) | 2 (2)
Bardycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bibasilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bibasilar opacities (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral basilar crackles (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bilateral Basilar Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin) (Skin and subcutaneous tissue disorders) | 1 (1)
Blurry Vision (Nervous system disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Brown Urine (Renal and urinary disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Chills (Nervous system disorders) | 7 (7)
Cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Cold right hand finger tips (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Nervous system disorders) | 3 (3)
Conjunctiva erythema (Vascular disorders) | 1 (1)
Conjunctival hemorrhage (Vascular disorders) | 1 (1)
Conjunctivitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Coughs (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine elevated (Endocrine disorders) | 1 (1)
Dark purple feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased breath sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep Vein Thrombosis, Left Arm (Vascular disorders) | 1 (1)
Dermatitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetes (Endocrine disorders) | 1 (1)
Diaphoresis (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Diffuse tenderness to deep palpation (Musculoskeletal and connective tissue disorders) | 1 (1)
Distal feet pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Distress (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Drowsy (Nervous system disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Edema (extremities) (Vascular disorders) | 2 (2)
Edema: head and neck, periorbital (Vascular disorders) | 2 (2)
Edema-limbs lower (Vascular disorders) | 4 (4)
Edema-limbs upper (Vascular disorders) | 2 (2)
Electrocytes Imbalance (Vascular disorders) | 1 (1)
Elevated alanine aminotransferase (Vascular disorders) | 2 (2)
Elevated aspartate transaminase (Vascular disorders) | 3 (3)
Elevated blood pressure (Vascular disorders) | 1 (1)
Enterococcus faecium (Endocrine disorders) | 1 (1)
Erythematous Joint, Left Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Erythematous Nodule (Vascular disorders) | 1 (1)
Facial Edema (Vascular disorders) | 1 (1)
Fatigue (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Febrile (Nervous system disorders) | 1 (1)
Fever (Nervous system disorders) | 11 (11)
Fingertip Numbness (Musculoskeletal and connective tissue disorders) | 1 (1)
Fluid overload (Endocrine disorders) | 1 (1)
Flushing arms/neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric extension (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Generalized Skin Erythema (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematomas (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hemorrhoidal Pain (Vascular disorders) | 1 (1)
Hemorrhoids (Vascular disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperbilirubinemia (Endocrine disorders) | 7 (7)
Hyperglycemia (Endocrine disorders) | 7 (7)
Hypermagnesemia (Endocrine disorders) | 2 (2)
Hypernatremia (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)
Hyphosphatemia (Vascular disorders) | 3 (3)
Hypoalbuminemia (Skin and subcutaneous tissue disorders) | 8 (8)
Hypocalcemia (Vascular disorders) | 8 (8)
Hypokalemia (Vascular disorders) | 9 (9)
Hypomagnesemia (Vascular disorders) | 5 (5)
Hyponatremia (Vascular disorders) | 10 (10)
Hypotension (Vascular disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infected peripherally inserted central catheter (PICC) Site (Musculoskeletal and connective tissue disorders) | 1 (1)
International Normalized Ratio Creased (Vascular disorders) | 2 (2)
Internal Bleeding (Vascular disorders) | 1 (1)
Irregular heart rhythm/rate (Cardiac disorders) | 2 (2)
Ischemia (Cardiac disorders) | 1 (1)
Labored breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Ankle Edema (Cardiac disorders) | 1 (1)
Left arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 5 (5)
Low aspartate aminotransferase (Cardiac disorders) | 1 (1)
Low auto platelet count (Cardiac disorders) | 2 (2)
Lymphedema Lower Extremity (Endocrine disorders) | 1 (1)
Lymphocyte count decreased (Cardiac disorders) | 1 (1)
Lymphopenia (Cardiac disorders) | 7 (7)
Macular rash (Musculoskeletal and connective tissue disorders) | 3 (3)
Mixed bilirubinemia (Endocrine disorders) | 1 (1)
Wall thickening of the cecum & ascending (Gastrointestinal disorders) | 1 (1)
Monocyte decrease (Cardiac disorders) | 1 (1)
Mood alteration: Anxiety (Nervous system disorders) | 3 (3)
Mottled lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Nervous system disorders) | 9 (9)
Neutropenia (Cardiac disorders) | 10 (10)
Neutrophil Count decreased (Cardiac disorders) | 2 (2)
Neutrophil Count increased (Cardiac disorders) | 1 (1)
No palpable dorsalis pedis pulses (Cardiac disorders) | 1 (1)
Numbing of bilateral feet (Nervous system disorders) | 1 (1)
Numbness/tingling in bilateral feet (Nervous system disorders) | 1 (1)
Oral candidiasis (Gastrointestinal disorders) | 1 (1)
Pain - Headache (Nervous system disorders) | 3 (3)
Pain - Other, Peripherally Inserted Central Catheter (PICC) line site (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain- Abdominal (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain at sacrum (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)
Pancytopenia (Cardiac disorders) | 3 (3)
Paranoia (Psychiatric disorders) | 1 (1)
Peripheral digital ischemia (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Positive Blood Cultures (Cardiac disorders) | 1 (1)
Positive for Gallops (Cardiac disorders) | 1 (1)
Preicardial effusion (Cardiac disorders) | 1 (1)
Pressor-related ischemia (Cardiac disorders) | 1 (1)
Prostatitis (Renal and urinary disorders) | 1 (1)
Proteinuria (Endocrine disorders) | 1 (1)
Pruritis (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Pulmonary crackles (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulseless electrical activity (Nervous system disorders) | 1 (1)
Pulseless legs (Nervous system disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales and Crackles, Bilat w Bases (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Musculoskeletal and connective tissue disorders) | 11 (11)
Rash on Trunk (Musculoskeletal and connective tissue disorders) | 2 (2)
Rash, Back, Abdomen (Musculoskeletal and connective tissue disorders) | 2 (2)
Rash, Facial (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Rectal Abscess (Gastrointestinal disorders) | 1 (1)
Renal Failure, acute (Endocrine disorders) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right lower lobe patchy opacification (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rigors (Nervous system disorders) | 10 (10)
Ringing in the ears (Nervous system disorders) | 1 (1)
Scrotal Swelling (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Shortness of breathe (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin Desquamation (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin Erythema, Back and Torso (Musculoskeletal and connective tissue disorders) | 1 (1)
Sloughing of skin in bilateral buttocks (Musculoskeletal and connective tissue disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Sputum (Gastrointestinal disorders) | 1 (1)
Stomach Gas (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Subconjunctival hemorrhage in both eyes (Cardiac disorders) | 1 (1)
Subcutaneous edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Subsegmental atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sweat (Musculoskeletal and connective tissue disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
Tachypenia (Cardiac disorders) | 1 (1)
Tachypneic (Cardiac disorders) | 1 (1)
Thrombocytopenia (Cardiac disorders) | 1 (1)
Upper gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
Upset Stomach (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 11 (11)
Uveitis (Musculoskeletal and connective tissue disorders) | 4 (4)
Visual hallucinations (Nervous system disorders) | 1 (1)
Vitiligo (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White Blood Cell decreased (Cardiac disorders) | 1 (1)
Tachypenic (Cardiac disorders) | 4 (4)
Insomnia (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT00910650/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT00910650/ICF_001.pdf